CLINICAL TRIAL: NCT04821128
Title: An Evaluation of the Radio/Pathological Correlation of Depth Of Invasion for Oral Squamous Cell Carcinoma, a Retrospective Study in a University Hospital in Lyon
Brief Title: Radio/Pathological Evaluation of Tongue Cancer Infiltration
Acronym: RaP E ToC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 242
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Oral Squamous; Cell Carcinoma
Keywords: DOI; Infiltration; Oral cavity cancer; OSCC; Tongue cancer; CT scanner
MeSH Terms: conditions — Mouth Neoplasms; Tongue Neoplasms | interventions — X-Rays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who improved surgical treatment for oral cavity cancer: T1 T2 and T3 OSCC tumor, patients who have a recent evaluation cervico thoracic scanner in their medical files.
  Interventions: Other: Radiologic and pathological review.

INTERVENTIONS:
Other: Radiologic and pathological review. — We will analyse the pre operative scannographic and MRI (if available) images, and the post operative pathological analyses.
  The scanners will be reviewed by 2 well trained clinicians (one head and neck radiologist and one head and neck surgeon).
  Then we will analyse the correlation between the radiological and the pathological analysis.

SUMMARY:
The aim of the study is to assess the good correlation and prediction of the DOI for the post-operative pathological results and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* patients chirurgically treated for an OSCC
* T1 T2 T3
* CT scanner in their medical file

Exclusion Criteria:

* T4
* R+ résection
* Artefacts on CT scanner

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population will include all the patients chirurgically treated for an OSCC for 2014 to 2019, who have a pre operativ scanner at least in their medical file.
  We will exclude the T4, the patients with very artefacted exams, and those with R+ resections.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2021-05-27 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the measure of the correlation of the depth of invasion on the radiological pre operative images and of the pathological analyses on the resection piece. | The outcome will be measured at the inclusion of the patient in the current study.
  With a Bland Altman analysis we will assess the good correlation between the pre and post operatory mesures of the depth of invasion in the oral squamous cell carcioma

CONTACTS AND LOCATIONS:
Locations (1):
- Croix rousse hospital, Lyon, France